CLINICAL TRIAL: NCT04391725
Title: Healing Following Use Of Injectable Platelet Rich Fibrin With Collagen During Surgery In Through And Through Periapical Lesions
Brief Title: Guided Tissue Regeneration in Healing of Through and Through Periapical Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Arpitha CM
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2019-12

CONDITIONS: Periapical Lesion
MeSH Terms: interventions — Guided Tissue Regeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periapical surgery with guided tissue regeneration (Experimental): Patients with through and through periapical lesion will undergo periapical surgery and the defect is filled with mixture of iPRF and type 1 collagen granules before flap closure.
  Interventions: Procedure: Periapical surgery with guided tissue regeneration
- Periapical surgery without any guided tissue regeneration (Active Comparator): Patients with through and through periapical lesion will undergo periapical surgery and flap closure done.
  Interventions: Procedure: Periapical surgery without anyguided tissue regeneration

INTERVENTIONS:
Procedure: Periapical surgery with guided tissue regeneration — periapical surgery will be done followed by placement of mixture of iPRF and type 1 collagen granules
  Arms: Periapical surgery with guided tissue regeneration
Procedure: Periapical surgery without anyguided tissue regeneration — periapical surgery will be done followed by flap closure
  Arms: Periapical surgery without any guided tissue regeneration

SUMMARY:
Aim of this study is to evaluate the effect of i-PRF in the healing of through and through periapical lesion after periradicular surgery

DETAILED DESCRIPTION:
Detailed patient examination will be carried out and those satisfying inclusion criteria will be enrolled in the study. Written informed consent will be obtained and patients will be randomly allocated to two groups. Entire surgical procedure will be carried out by single operator. After complete elevation of the flap, debridement (periradicular curettage -enucleation) of the bony lesion will be performed. 3 mm root-tip resection will be performed and root end cavity will be prepared using an ultrasonic diamond-coated retrotip. Root end filling will be done with mineral trioxide aggregate (MTA). In test group The i-PRF will be produced and incorporated with collagen will be used to fill into the defect. In the control group, no guided tissue regeneration technique will be used. Flap will be re-positioned and sutured using nonabsorbable 4-0 silk sutures.Sutures will be removed 4-7 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 16-55 years with a clinical & radiographic diagnosis of through and through periradicular lesion using CBCT
* Negative response to sensitivity tests with radiographic evidence of periapical radiolucency.
* Failed previous root canal treatment primary or secondary with purulent discharge and radiographic evidence of periapical pathology.
* The teeth must have adequate final restoration with no clinical evidence of coronal leakage.

Exclusion Criteria:

* Unrestorable tooth.
* Fractured / perforated tooth.
* Systemic diseases contraindicating surgical procedures or with potential to affect healing.
* Teeth with deep pockets.
* Patient requiring antibiotic premedication.
* Patients with history of antibiotic use in last 3 months.
* Smokers

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-12-11 (Estimated); Study Completion 2021-04-11 (Estimated)

PRIMARY OUTCOMES:
change from baseline in periapical radiolucency at 12 months | baseline to 12 months
  2 blinded caliberated operators will score the periapical radiolucency at baseline and 12 month with following scoring scores for 2D healing Score 1 - Complete healing, defined by re-establishment of the lamina dura Score 2 - Incomplete healing (scar tissue) Score 3 - Uncertain healing Score 4 - Unsatisfactory healing (failure)
  scores for 3D healing Score 1 - Complete healing Score 2 - Limited healing Score 3 - Uncertain healing Score 4 - Unsatisfactory healing

SECONDARY OUTCOMES:
change in Quality of life from baseline to 7 days | postoperative Day 1 to day 7
  caliberated operator will score the quality of life questionnaire in patients following surgical endodontic treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sanjay Tewari, Rohtak, Haryana, India

REFERENCES:
- [Derived] M A, S T, P S, A G. Efficacy of mixture of injectable-platelet-rich fibrin and type-1 collagen particles on the closure of through-and-through periapical bone defects: A randomized controlled trial. Int Endod J. 2023 Oct;56(10):1197-1211. doi: 10.1111/iej.13954. Epub 2023 Jul 17. PMID 37418583